CLINICAL TRIAL: NCT05151965
Title: Return to Sport and Functional Performance Following Surgical Intervention for Anterior Glenohumeral Instability (AGHI)
Brief Title: Return to Sport and Functional Performance Following Surgical Intervention for Anterior Glenohumeral Instability
Status: Recruiting | Type: Observational
Sponsor: Panam Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: B2021:094
Record Dates: First submitted 2021-11-26; First posted 2021-12-09 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Anterior Shoulder Dislocation; Anterior Shoulder Instability
Keywords: Bankart repair; Remplissage; Latarjet Coracoid Transfer; Return to sport

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bankart Repair and Remplissage: Patients will undergo a standard arthroscopic anterior labral repair with a minimum of 3 suture anchors, followed by remplissage with 1 or 2 anchors, at the discretion of the treating surgeon.
  Interventions: Procedure: Bankart Repair and Remplissage
- Latarjet Coracoid Transfer: Patients will undergo a Latarjet coracoid transfer through a deltopectoral approach and horizontal split in the subscapularis at the superior 2/3, inferior 1/3 junction. The coracoid process will be oriented in the conventional manner, with the inferior surface against the glenoid vault, secured with two cannulated screws
  Interventions: Procedure: Latarjet Coracoid Transfer

INTERVENTIONS:
Procedure: Bankart Repair and Remplissage — Arthroscopic Bankart repair with a minimum of 3 anchors
  1 or 2 anchor Remplissage subsequently performed with percutaneous anchor insertion in the base of the Hill-Sachs defect, and sutures passed in a horizontal mattress configuration 1 cm apart, tied in the subacromial space.
  Groups: Bankart Repair and Remplissage
Procedure: Latarjet Coracoid Transfer — Coracoid transfer performed via deltopectoral approach with horizontal subscapularis split. Graft placed in the conventional orientation, secured with 2 screws, ensuring the graft is not lateral to the glenoid rim.
  Groups: Latarjet Coracoid Transfer

SUMMARY:
The purpose of this prospective cohort study is to compare patient-reported, clinical, and functional outcomes in patients who have elected to have either the Bankart with Remplissage or Latarjet procedure for the treatment of anterior glenohumeral instability (AGHI) up to 24-months postoperative.

DETAILED DESCRIPTION:
The purpose of this prospective cohort study is to compare patient-reported, clinical, and functional outcomes in patients who have elected to have either the Bankart with Remplissage or Latarjet procedure for the treatment of AGHI up to 24-months postoperative. A secondary objective aims to address rates of return to sport (RTS) and performance in an RTS assessment in athletic patients with anterior glenohumeral instability (AGHI) who elect to undergo either surgical intervention until 24-months postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 50 years
* Documented reduction of anterior shoulder dislocation
* Patient has suffered two or more dislocations of the study shoulder
* Physical examination elicits unwanted glenohumeral translation with reproduction of symptoms
* Glenoid bone loss defined on CT (or MRI) using standardized and reproducible best-fit circle techniques < 25%
* Able to benefit from surgical intervention

Exclusion Criteria:

* Glenoid defect in the affected shoulder ≥ 25% of the AP diameter of the glenoid
* Previous surgery on affected shoulder (ANY type of shoulder surgery)
* Significant shoulder comorbidities including osteoarthritis or other shoulder conditions including multi-directional instability
* Participant is involved in litigation or a workplace insurance claim (i.e., WCB).
* Confirmed connective tissue disorder (i.e., Ehlers-Danlos, Marfans)
* Beighton hypermobility score of >6
* Active joint or systemic infection, significant muscle paralysis, rotator cuff tear arthropathy, Charcot's arthropathy, significant medical comorbidity that could alter the effectiveness of the surgical intervention (e.g., Cervical radiculopathy, polymyalgia rheumatica)
* Major medical illness (life expectancy less than 1 year) or unacceptably high operative risk
* Epilepsy
* Any condition that precludes informed consent (i.e. psychiatric illness)
* Unable to speak or read English/French
* Unable or unwilling to be followed for 2 years or complete functional testing

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults aged 18 - 50 years who have documented reduction of anterior shoulder dislocation. The participant has suffered two or more dislocations of the study shoulder, and the physical examination elicits unwanted glenohumeral translation with reproduction of symptoms. The participant has glenoid bone loss defined on CT (or MRI) using standardized and reproducible best-fit circle techniques < 25%, and would benefit from surgical intervention.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Western Ontario Shoulder Instability Index (WOSI) | 24 months
  Is a disease specific, quality of life patient reported outcome measures (PROMS) for patients with shoulder instability. Patients use visual analog scales (VAS) to rate physical symptoms and impacts of the condition/treatment on sports/recreation/work, lifestyle, and emotions.
Shoulder dislocation and recurrence | 24 months
  Dislocation requiring reduction by a physician (ED) or surgery. Dislocations will be identified in two ways: 1) if the patient seeks treatment from the surgeon, the surgeon will notify the research coordinator who will document it accordingly, or 2) at each research postoperative examination, the research staff will ask patients if they experienced a dislocation or subluxation. These will be considered alongside the definition of recurrence from Kasik et al. that also includes subluxation, or positive findings during physical examination for shoulder instability (apprehension).
Surgical complications, re-operations and revision surgeries | 24 months
  Surgical complications will be documented at the time of surgery and at each postoperative interval. A surgical complication is defined as any undesirable, unintended and direct result of an operation affecting the patient that would not have occurred had the operation gone well as could reasonably be hoped (Sokol and Wilson, 2008) (i.e., infection, dislocation, neurological injury, and fracture (including periprosthetic and acromial fracture).
  Revision surgery and re-operations will be documented, including the reason for failure, date of revision/reoperation, and the procedure performed. Revision is defined as a change of an original component (partial or complete replacement). Re-operation is defined as any surgical procedure other than a revision.

SECONDARY OUTCOMES:
Isokinetic Internal and External Rotation | 24 months
  Internal and external rotation strength will be determined with an isokinetic dynamometer (Biodex Medical Systems, Shirley, NY, USA). With the arm in 90 degrees shoulder abduction and elbow flexion and positioned in the scapular plane, patients will complete coupled concentric and eccentric shoulder internal and external rotation within a 90 degrees range of motion (-40 degrees internal rotation to 50 degrees external rotations). Three maximal effort (instructed to contract as hard and as fast as they can) repetitions will be completed at velocities of 60 and 180 degrees per second, with one-minute rest between testing speeds. Average peak torque of the three repetitions will be recorded for both IR and ER.
Athletic Shoulder (ASH) Test | 24 months
  The patient Is positioned prone with a foam block in place to support their forehand. The test is completed in three positions termed "I", with the arm positioned in 180 degrees of shoulder flexion, "Y, with the arm positioned in 135 degrees of shoulder abduction, and "T", with the arm positioned in 90 degrees of abduction. In each position, the palm of the hand rests on a force plate (AMTI, MA, USA). The patient will complete a warm-up of two submaximal attempts in each position to 80-90% maximal effort, then three maximal effort trials for each limb in each test position (I, Y, T), with 20 seconds rest between repetitions. For each repetition, subjects will be instructed to push against the plate as hard and as fast as possible for three seconds. Peak and mean force across the three attempts and positions will be recorded.
Seated medicine ball toss | 24 months
  The patient will start the test in the seated position with the legs extended in front of their body, and the head, shoulders and back firmly against a wall. They will then attempt a "chest pass" by throwing a 10 lbs. medicine ball as far as they can. Four trials will be completed with 30 sec rest between each trial. Maximum distance will be recorded and averaged, once adjusted for arm length (distance of the ball from the wall with the arm held at 90 degrees of flexion and full elbow extension).
Posterior Shoulder Endurance Test | 24 months
  The patient starts positioned in prone towards one edge of a plinth, with the arm held in 90o shoulder flexion, perpendicular to the floor. Holding a weight of 2% of total body weight, the patient will attempt to raise the weight to 90 degrees of horizontal abduction, holding for one second at this position before returning to the starting position (tempo of 30 bpm). The test is terminated when the patient is fatigued as indicated by 1) the inability to hold the mid position for one second and 2) using compensatory movements of the torso, or patient request to terminate.
Plyometric Push up | 24 months
  Participants will start in a push up position with each hand extended in front of the shoulders and positioned on an individual force plate. When cued, the participant will lower their body to the ground by flexing at the elbow until their sternum is 3 cm from the floor. They will then forcefully extend at the elbow and propel their body into the air above the plate. During landing, the subjects will be instructed to reduce the impact as much as possible and continue for two additional repetitions. Three repetitions will be completed. Peak ground reaction forces during impact, peak rate of force development (RFD) during the concentric phase will be averaged from the three repetitions and expressed as a limb symmetry index (injured/uninjured * 100%).
Single arm seated shot put | 24 months
  The patient will start seated in an 18" chair without arm rests, with the legs positioned in front of their body, extended to rest straight onto an additional chair. The non-throwing arm will be placed across the chest, with a strap placed diagonally around the upper body to secure the subject to the chair. The patient will "put" (like shot put), and not "throw" (like baseball) the 6 lb. ball from shoulder height for maximal distance. Three maximal effort attempts will be recorded after a graded warm-up of four "puts" at 25, 50, 75 and 100% estimated effort. Thirty seconds rest will be provided between maximal attempts.

OTHER OUTCOMES:
American Shoulder and Elbow Surgeons Standardized Shoulder Assessment form (ASES) | 24 months
  The ASES is a patient-reported upper extremity functional assessment tool and is scored out of a maximum 100 points, that represents maximum function and no pain.
Single Assessment Numeric Evaluation (SANE) score | 24 months
  Is a single question that asks patients to rate their affected shoulder as a percentage of normal, "How would you rate your affected shoulder today as a percentage of normal (0% to 100% scale with 100% being normal)?"
EuroQol-5D (EQ-5D) + Visual Analog Scale (VAS) | 24 months
  The EQ-5D is a PROM used to document overall wellness across five dimensions including mobility, self-care, usual activities, pain and anxiety/depression. A single value is calculated to represent the patients' health state relative to a specific population. The VAS asks participants: We would like you to indicate on this scale how good or bad your own health is TODAY, in your opinion. 100 means the best health you can imagine. 0 means worst health you can imagine.
Shoulder activity scale (SAS) | 24 months
  A patient reported outcome measure (PROM) where patients categorize the frequency (i.e. never, once a month, once a week, more than once a week, and daily) of certain activities of the upper extremity (i.e. carrying objects 8 lbs. or heavier by hand) and also identify whether they participate in either contact or overhead sports including the level of participation.
Postoperative Pain and Medication Use | 3 weeks
  Postoperative pain will be self-reported on a 100mm visual analogue scale (VAS) in a logbook. Medication type and quantity will also be documented. The Postoperative Pain and Medication Logbook has been previously used by the authors in an ACL population.
Subjective Patient Outcome for Return to Sports (SPORTS) | 24 months
  Evaluates the ability of an athlete to resume their sport at-pre-injury level of training or performance, and whether each is possible without or despite pain. Scored on a 10-point scale, where an inability to return to the same sport is scored as "0" and unlimited effort and performance without pain is a "10".
Shoulder Instability Return to Sport (SIRSI) | 24 months
  PROM of psychological readiness to return-to-sport (RTS), adapted from the previously validated ACL-RSI, that may highlight clinically important differences in patient's perceptions relative to RTS between the two procedures. The SIRSI asks participants 12 questions where they rate on a 10-point scale; "0" is not confident at all, and "10" is fully confident.
Waterloo Handedness Questionnaire (WHQ) | 24 months
  A series of 39 questions used to establish limb dominance, where questions 1-36 ask the participant to indicate their hand preference for the following activities by circling the appropriate response. If they always (i.e. 95% or more of the time) use one hand to perform the described activity, circle Ra or La (for right always or left always). If they usually (i.e. about 75% of the time) use one hand circle Ru or Lu, as appropriate. If they use both hands equally often (i.e. you use each hand about 50% of the time), circle Eq. Questions 37-39 are 'Yes" or "No" answers.
Closed Kinetic Chain Upper Extremity Stability Test | 24 months
  The patient assumes a standard push-up position with the middle of the hands positioned on a 1.5" piece of athletic tape, with 36" between each piece of tape. The patient then alternates lifting each hand to touch the opposite hand/tape as many times as possible within 15 seconds. Three trials will be completed and averaged. Thirty seconds rest will be provided between trials.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Ogborn, PhD, Principal Investigator — Pan Am Clinic
Locations (1):
- Pan Am Clinic, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers.